CLINICAL TRIAL: NCT05505240
Title: Influence of Ambient Temperature on Resting Energy Expenditure of Metabolically Healthy Men and Women
Brief Title: Influence of Ambient Temperature on Resting Energy Expenditure of Healthy Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bonn (Other)
Collaborators: DLR German Aerospace Center (Other)
Responsible Party: Principal Investigator, Prof. Dr. Sarah Egert, Prof. PhD, University of Bonn
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: TempRMR
Record Dates: First submitted 2022-08-15; First posted 2022-08-17 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Resting Energy Expenditure
Keywords: Resting energy expenditure; Resting metabolic rate; Ambient temperature; Environmental temperature

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Cold temperature (Experimental): 18°C
  Interventions: Other: Respiratory analysis at cold temperature
- Room temperature (Experimental): 22°C
  Interventions: Other: Respiratory analysis at room temperature
- Thermoneutral temperature (Experimental): 28°C
  Interventions: Other: Respiratory analysis at thermoneutral temperature
- Hot temperature (Experimental): 38°C
  Interventions: Other: Respiratory analysis at hot temperature

INTERVENTIONS:
Other: Respiratory analysis at cold temperature — Respiratory analysis at an ambient temperature of 18°C
  Arms: Cold temperature
Other: Respiratory analysis at room temperature — Respiratory analysis at an ambient temperature of 22°C
  Arms: Room temperature
Other: Respiratory analysis at thermoneutral temperature — Respiratory analysis at an ambient temperature of 28°C
  Arms: Thermoneutral temperature
Other: Respiratory analysis at hot temperature — Respiratory analysis at an ambient temperature of 38°C
  Arms: Hot temperature

SUMMARY:
The aim of this study is to investigate the influence of four different ambient temperatures (18, 22, 28, 38°C) on the resting energy expenditure of healthy adults by respiratory gas analysis. It is assumed that the resting energy expenditure is higher at 18°C and 38°C than at the temperatures in between.

DETAILED DESCRIPTION:
In a crossover-design, 32 healthy men and women participate in four interventions. Each intervention includes a measurement of the resting energy expenditure by respiratory gas analysis at a different ambient temperature (18,22, 28 and 38°C). During this time body core- and surface temperature are assessed, as well as body composition via bioelectrical impedance analysis. For each participant the four individual study days take place in a randomized order on consecutive weekdays within a week.

ELIGIBILITY:
Inclusion Criteria

* BMI: 18,5 - 24,9 kg/m2
* metabolically healthy

Exclusion Criteria

* smoking
* low or high blood pressure
* dyslipidemia
* insulin resistance or diabetes mellitus type 1 or type 2
* gastrointestinal diseases (e.g. food intolerances or allergies)
* liver, kidney and/or thyroid diseases
* hepatitis B or C, HIV Infection
* chronic inflammatory diseases
* disordered eating
* psychological diseases
* alcohol and/or drug abuse
* use of medication
* pregnancy or lactating
* participation in another intervention study
* women: irregular menstrual cycle
* more than 6 h of sports per week

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2022-11-21 (Actual); Primary Completion 2023-04-06 (Actual); Study Completion 2023-04-06 (Actual)

PRIMARY OUTCOMES:
Resting Energy Expenditure | 20 minutes
  Volume of inhaled oxygen (VO2) in L/min and exhaled carbon dioxide (VCO2) in L/min

SECONDARY OUTCOMES:
Body core temperature | 20 minutes
  Body core temperature: assessed every ten seconds during respiratory analysis (°C)
Body surface temperature | 20 minutes
  Body surface temperature: assessed every ten seconds during respiratory analysis (°C)
Body composition | 5 minutes (after respiratory analysis)
  assessed daily via bioelectrical impedance analysis after respiratory analysis (FFM (kg), FM (kg))
Blood pressure | 10 minutes (at beginning of study day)
  assessed daily before respiratory analysis (mmHg)

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Egert, Prof. PhD, Principal Investigator — University of Bonn
Locations (1):
- University of Bonn, Bonn, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Henkel S, Frings-Meuthen P, Diekmann C, Coenen M, Stoffel-Wagner B, Nemeth R, Pesta D, Egert S. Influence of Ambient Temperature on Resting Energy Expenditure in Metabolically Healthy Males and Females. J Nutr. 2025 Mar;155(3):862-870. doi: 10.1016/j.tjnut.2025.01.013. Epub 2025 Jan 13. PMID 39814140